CLINICAL TRIAL: NCT06122181
Title: A Randomized, Double-blind, Placebo-controlled Phase Ib Clinical Study to Evaluate the Safety, Tolerability and Pharmacokinetics Characteristics of HS-10384 in Chinese Postmenopausal Women
Brief Title: Study of HS-10384 in Participants of Chinese Postmenopausal Women
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Hansoh BioMedical R&D Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: HS-10384-102
Record Dates: First submitted 2023-11-03; First posted 2023-11-08 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Vasomotor Symptoms
Keywords: HS-10384; multiple ascending dose; postmenopausal women

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HS-10384 (Experimental): Multiple ascending doses of HS-10384 orally
  Interventions: Drug: HS-10384 tablets
- Placebo (Placebo Comparator): Multiple ascending doses of HS-10384 placebo orally
  Interventions: Drug: HS-10384-matched placebo tablets

INTERVENTIONS:
Drug: HS-10384 tablets — Multiple dosing of HS-10384 orally in a fasting state
  Arms: HS-10384
Drug: HS-10384-matched placebo tablets — Multiple dosing of HS-10384-matched placebo orally in a fasting state
  Arms: Placebo

SUMMARY:
A randomized, double-blind, placebo-controlled phase Ib clinical study to evaluate the safety, tolerability and pharmacokinetics characteristics of HS-10384 in Chinese postmenopausal women.

DETAILED DESCRIPTION:
Phase Ib is consisted with 3~4 multiple ascending doses.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects should fully understand the content, process and possible adverse reactions of the study, and voluntarily sign the informed consent form;
2. Age between 40 and 65 years old (including the critical value);
3. The body mass index (BMI=body weight [kg]/height2 [m2]) at screening is 19~28 kg/m2 (including the critical value of 19), and the weight is ≥ 40 kg;
4. Subjects are postmenopausal women at screening as qualified by any of the following criteria: spontaneous amenorrhea ≥ 12 months, or spontaneous amenorrhea ≥ 6 months and FSH>40 IU/L (without other obvious pathological or physiological reasonsbefore screening), or documented surgical sterilization (such as hysterectomy, bilateral salpingectomy or bilateral oophorectomy, etc.);
5. From 48 hours before taking drug to the end of the study, subjects should avoid taking tobacco products, alcohol and other foods or drinks that might affect drug metabolism (such as coffee, tea, cola or other caffeinated drinks);
6. The blood pregnancy test of female subjects at baseline period is negative.

Exclusion Criteria:

1. Participants with disease history of uterine bleeding, uterine ovarian tumor, pituitary tumor, or other diseases evaluated by the principal investigator as not suitable for this study;
2. Have a history of migraine within 3 months before screening;
3. Participants with clinically significant diseases (such as neuropsychiatric system, cardiovascular system, urinary system, digestive system, respiratory system, skeletal muscle system, endocrine and metabolic system, blood system, skin disease, immune system, tumor, etc.) were evaluated by the researcher as not suitable for this study;
4. Within 2 weeks before screening, participants have suffered from VMS that inducing the interrupt of daily activities;
5. Within 30 days before taking drug, participants have taken hormonal treatment or other therapy due to VMS;
6. Within 4 weeks or 5 half-lives (whichever is longer) before screening, and during the whole study period, it is expected to take any medicine and health care products, including prescription drugs, immunomodulator or Chinese herbal medicine, etc.;
7. Within 3 months before screening, participants have taken hormonal contraceptive;
8. Participants have participated in any clinical study or taken study drugs within 3 months before screening;

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2023-11-12 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
The incidence and severity of adverse events (AE), serious adverse events (SAE) and adverse events leading to withdrawal from the trial and the correlation with the investigational drug; | Day 1 to Day 21
Number of participants with clinical laboratory abnormalities | Day 1 to Day 21
  Clinical laboratory tests include blood routine, blood biochemistry, coagulation function, urine routine, thyroid function,etc.
Number of participants with abnormalities of vital signs | Day 1 to Day 21
Number of participants with abnormalities of physical examination | Day 1 to Day 21

SECONDARY OUTCOMES:
Cmax | Day 1 to Day 13
  Maximum plasma concentration
Tmax | Day 1 to Day 13
  Time to Cmax
AUC0-24 | Day 1 to Day 13
  Area under plasma concentration-time curve from time 0 to 24 h
Css,max | Day 14 to Day 21
  Maximum plasma concentration at steady state
Tss,max | Day 14 to Day 21
  Time to Cmax at steady state
Css,min | Day 14 to Day 21
  Minimum plasma concentration at steady state
AUCss | Day 14 to Day 21
  Area under plasma concentration-time curve in one dosing interval at steady state
RAC | Day 14 to Day 21
  Degree of accumulation after multiple doses
Luteinizing hormone changes from baseline | Day 1 to Day 21

CONTACTS AND LOCATIONS:
Overall Officials: Rong Li, PhD, Principal Investigator — Peking University Third Hospital; Dongyang Liu, Principal Investigator — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China